CLINICAL TRIAL: NCT02001467
Title: The Effects of Simulation-based Ultrasound Training on Continuity of Care in Managing Pre-mature Onset of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Martin G. Tolsgaard, MD, PhD, postdoctoral fellow, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-4-2013-FSP 10; H-4-2013-FSP 10 (Other: Regional Ethical Committee of the Capital Region, Denmark)
Record Dates: First submitted 2013-11-21; First posted 2013-12-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Continuity of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simulation-based training (Active Comparator): Simulation-based training to an expert criterion followed by clinical training until proficiency and certification.
  Interventions: Other: Simulation-based training
- Control (No Intervention): No training is provided the control group participants.

INTERVENTIONS:
Other: Simulation-based training
  Other Names: Simulation-based training on a high-fidelity ultrasound simulator (Scantrainer, Medaphor) and subsequently on a low-fidelity mannequin (BluePhantom, CAE).
  Arms: Simulation-based training

SUMMARY:
Simulation-based training lead to improvements in learning compared to no intervention but little is known of the effects on organizational improvements that are relevant to patient care. This study focused on the effects of training midwives in performing cervical ultrasound scans on continuity of care when managing pregnant women with symptoms of premature onset of labor. Our hypothesis is that simulation-based training can be used to decrease the number of shifts in primary responsible health care practitioner as midwives that are trained in cervical ultrasound scans may manage the patient encounter without engaging a second practitioner (i.e. an obstetrician).

DETAILED DESCRIPTION:
Pregnant women with symptoms of premature onset of labor are typically managed by midwives and obstetricians but shifts in responsibility in patient care may result in lack of continuity of care. This may, in turn, result in threats to patient safety and delays in initiation of treatment due to long wait times.

This study examined the effects of simulation-based ultrasound training on the management of women with symptoms of pre-mature onset of labor. 12 midwives were randomized to simulation-based ultrasound training focusing on cervical assessment or no training (controls). The midwives in the intervention group were trained to an expert criterion on a high-fidelity transvaginal ultrasound simulator. Once this level was attained, they continued clinical training until proficiency in performing cervical scans independently. Proficiency was determined using a previously validated assessment instrument (the Objective Structured Assessment of Ultrasound Skills) and by sending in pictures for the Fetal Medicine Foundation certification programme.

The number of responsible health care practitioners providing care for pregnant women with acute onset of symptoms of premature onset of labor is registered along with time from arrival at the hospital to medical assessment and treatment is commenced. Differences between patients treated by the two groups of midwives are compared over a period of 6 months. During this period all patients with symptoms of premature onset of labor are included, of which only a small proportion are admitted for further examinations and treatment. The vast majority are expected to be scheduled for ambulatory follow-up.

ELIGIBILITY:
Inclusion Criteria:

All midwives who are taking shift on the maternity ward

Exclusion Criteria:

Any prior ultrasound training and planned maternity leave.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Continuity of care | Patients will be followed untill discharge from the hospital, which is expected to be an average of 6 hours
  Continuity of care is evaluated by registering the number of health care practitioners involved in patient management.

SECONDARY OUTCOMES:
Wait times | An average of 6 hours is expected.
  Wait times for pregnant women with symptoms of premature onset of labor are registered and compared between the two groups of midwives, who are responsible for the initial patient care and -contact.

CONTACTS AND LOCATIONS:
Overall Officials: Martin G Tolsgaard, MD, PhD, Principal Investigator — CEKU
Locations (1):
- Nordsjællands Hospital, Hillerød, Capital Region, Denmark